CLINICAL TRIAL: NCT03683082
Title: Acute Effects of Oxygen Supplementation Among Pulmonary Arterial Hypertension Patients
Brief Title: Oxygen Treatment and Pulmonary Arterial Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: George Papanicolaou Hospital (Other)
Responsible Party: Principal Investigator, Afroditi Boutou, Consultant in Respiratory Medicine, George Papanicolaou Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 803/2018
Record Dates: First submitted 2018-09-20; First posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Air

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAH patients (Active Comparator): Supplementation of oxygen therapy (40% FiO2) during steady state cardiopulmonary exercise testing, via Venturi mask
  Interventions: Drug: Oxygen supplementation
- PAH patients (crossover) (Sham Comparator): Supplementation of medical air (sham oxygen) during steady state cardiopulmonary exercise testing, via Venturi mask
  Interventions: Drug: Sham O2 (medical air)

INTERVENTIONS:
Drug: Oxygen supplementation — 40% FiO2 via Venturi mask
  Arms: PAH patients
Drug: Sham O2 (medical air) — Medical air supplementation via Venturi mask
  Arms: PAH patients (crossover)

SUMMARY:
Pulmonary arterial hypertension (PAH) is a disease characterised with significant morbidity and poor prognosis. Dyspnoea and impaired exercise capacity are very common manifestations of the disease, and result in significant impairment of patients' quality of life. Although hypoxemia is common among subjects with PAH, published data on the effects of supplementary oxygen therapy on specific clinical outcomes among these patients are currently few, while the existing data on the potential benefits of oxygen supplementation to treat exercise-induced hypoxemia, in this patient population, are even more controversial. Based on the aforementioned, the purpose of this prospective, crossover clinical trial is to investigate the acute effects of supplemental oxygen administration on the: a) exercise capacity, b) severity of dyspnea, c) cerebral oxygenation, b) muscle oxygenation, and e) hemodynamic profile, as compared to delivery of medical air (sham oxygen), in a group of patients with PAH, during steady state cardiopulmonary exercise testing (CPET)

ELIGIBILITY:
Inclusion Criteria:

1. Group I PAH patients
2. Stable disease (no hospitalisation, disease deterioration or change in regular PAH medication during the last month)
3. Presence of exercise-induced hypoxemia

Exclusion Criteria:

1. Major contraindications for CPET conduction
2. Not providing informed consent -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-06-10 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Exercise duration | through study completion, an average of a year
  Exercise duration (minutes), while conducting steady state cardiopulmonary exercise testing until exhaustion

SECONDARY OUTCOMES:
Dyspnea | through study completion, an average of a year
  Maximum dyspnea assessed by Borg dyspnea scale, during steady state cardiopulmonary exercise testing
cerebral oxygenated hemoglobin | through study completion, an average of a year
  minimum value of cerebral oxygenated hemoglobin during steady state cardiopulmonary exercise testing
Cardiac output | through study completion an average of a year
  maximum cardiac output during steady state cardiopulmonary exercise testing
Fatigue | through study completion, an average of a year
  Maximum fatigue as assessed by Borg fatigue scale, during steady state cardiopulmonary exercise testing

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Pitsiou, MD, Ass Prof, Study Chair — "G. Papanikolaou" General Hospital, Thessaloniki, Greece
Locations (1):
- "G. Papanikolaou" General Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dipla K, Boutou AK, Markopoulou A, Papadopoulos S, Kritikou S, Pitsiou G, Stanopoulos I, Kioumis I, Zafeiridis A. Differences in cerebral oxygenation during exercise in patients with idiopathic pulmonary fibrosis with and without exertional hypoxemia: does exercise intensity matter? Pulmonology. 2023 May-Jun;29(3):221-229. doi: 10.1016/j.pulmoe.2021.06.006. Epub 2021 Jul 15. PMID 34274251
- [Derived] Boutou AK, Dipla K, Zafeiridis A, Markopoulou A, Papadopoulos S, Kritikou S, Panagiotidou E, Stanopoulos I, Pitsiou G. A randomized placebo-control trial of the acute effects of oxygen supplementation on exercise hemodynamics, autonomic modulation, and brain oxygenation in patients with pulmonary hypertension. Respir Physiol Neurobiol. 2021 Aug;290:103677. doi: 10.1016/j.resp.2021.103677. Epub 2021 May 3. PMID 33957299